CLINICAL TRIAL: NCT00314080
Title: An Outbreak of Botulism in Thailand: Clinical Manifestations and Management of Severe Respiratory Failure
Brief Title: Treatment of Survivors After Botulism Outbreak
Status: Completed | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Rajavithi Biomolecular Research Center (Other)
Other Study IDs: RVH_CER_001
Record Dates: First submitted 2006-03-30; First posted 2006-04-12 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2007-08

CONDITIONS: Respiratory Failure; Botulism
Keywords: Botulism; Botulinum anti-toxin; Repetitive nerve stimulation; Respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency; Botulism | interventions — Botulinum Antitoxin

INTERVENTIONS:
Drug: Botulinum AntiToxin
Procedure: neuro-electrophysiologic study, repetitive nerve stimulation
Procedure: Protocol early weaning ventilator after recovery of repetitive nerve stimulation and stable negative inspiratory pressure

SUMMARY:
Background. Northern Thailand's biggest botulism outbreak to date occurred on 14 March 2006 and affected 209 people. Of these, 42 developed respiratory failure, and 25 of those who developed respiratory failure were referred to 9 high facility hospitals for treatment of severe respiratory failure and autonomic nervous system involvement. Among these patients, we aimed to assess the relationship between the rate of ventilator dependence and the occurrence of treatment by day 4 versus day 6 after exposure to bamboo shoots (the source of the botulism outbreak), as well as the relationship between ventilator dependence and negative inspiratory pressure.

Methods. The investigators reviewed the circumstances and timing of symptoms following exposure. Mobile teams treated patients with botulinum antitoxin on day 4 or day 6 after exposure in Nan Hospital (Nan, Thailand). Eighteen patients (in 7 high facility hospitals) with severe respiratory failure received a low- and high-rate repetitive nerve stimulation test, and negative inspiratory pressure was measured.

ELIGIBILITY:
Inclusions:

* Ate the bamboo shoots in Banluang district, on March,14 2006
* Clinical of respiratory failure and need ventilator assistant
* Needed to referred to other hospital
* The staffs of referred hospital willing to participate in the Thai Botulism study group

Exclusion Criteria:

* Patients who did not eat bamboo shoots in Banluang district on March14,2006.
* No clinical of respiratory failure.
* Not referred to other hospital.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18
Dates: Start 2006-03; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Subsai Kongsaengdao, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

REFERENCES:
- [Background] World Health Organization .Botulism in Thailand: Epidemic and Pandemic Alert and Response (EPR). (Accessed March 22, 2006, at http://www.who.int/csr/don/2005_12_22/en/)
- [Background] P Wongwatcharapaiboon, L Thaikruea, and K Ungchusak et. al. Foodborne Botulism Associated With Home-Canned Bamboo Shoots,Thailand, 1998. ). (Accessed March 22, 2006, at http://www.cdc.gov/mmwr/preview/mmwrhtml/mm4821a1.htm)
- [Background] Swaddiwudhipong W, Wongwatcharapaiboon P. Foodborne botulism outbreaks following consumption of home-canned bamboo shoots in Northern Thailand. J Med Assoc Thai. 2000 Sep;83(9):1021-5. PMID 11075968
- [Background] Fernandez PS, Peck MW. A predictive model that describes the effect of prolonged heating at 70 to 90 degrees C and subsequent incubation at refrigeration temperatures on growth from spores and toxigenesis by nonproteolytic Clostridium botulinum in the presence of lysozyme. Appl Environ Microbiol. 1999 Aug;65(8):3449-57. doi: 10.1128/AEM.65.8.3449-3457.1999. PMID 10427033
- [Background] Zanon P, Pattis P, Pittscheider W, Roscia G, De Giorgi G, Sacco G, Votter K, Stockner I, De Giorgi F, Wiedermann CJ. Two cases of foodborne botulism with home-preserved asparagus. Anasthesiol Intensivmed Notfallmed Schmerzther. 2006 Mar;41(3):156-9. doi: 10.1055/s-2006-924967. PMID 16557441
- [Background] Jones RG, Corbel MJ, Sesardic D. A review of WHO International Standards for botulinum antitoxins. Biologicals. 2006 Sep;34(3):223-6. doi: 10.1016/j.biologicals.2005.11.009. Epub 2006 Feb 20. PMID 16490362
- [Background] Boyadjiev I, Leone M, Garnier F, Thomachot L, Martin C. [A case of type A botulism]. Ann Fr Anesth Reanim. 2005 Nov-Dec;24(11-12):1397-9. doi: 10.1016/j.annfar.2005.06.002. Epub 2005 Oct 26. French. PMID 16256299
- [Background] Sobel J. Botulism. Clin Infect Dis. 2005 Oct 15;41(8):1167-73. doi: 10.1086/444507. Epub 2005 Aug 29. PMID 16163636
- [Background] Agarwal AK, Goel A, Kohli A, Rohtagi A, Kumar R. Food-borne botulism. J Assoc Physicians India. 2004 Aug;52:677-8. No abstract available. PMID 15847370
- [Background] Sobel J, Tucker N, Sulka A, McLaughlin J, Maslanka S. Foodborne botulism in the United States, 1990-2000. Emerg Infect Dis. 2004 Sep;10(9):1606-11. doi: 10.3201/eid1009.030745. PMID 15498163
- [Result] Kongsaengdao S, Samintarapanya K, Rusmeechan S, Wongsa A, Pothirat C, Permpikul C, Pongpakdee S, Puavilai W, Kateruttanakul P, Phengtham U, Panjapornpon K, Janma J, Piyavechviratana K, Sithinamsuwan P, Deesomchok A, Tongyoo S, Vilaichone W, Boonyapisit K, Mayotarn S, Piya-Isragul B, Rattanaphon A, Intalapaporn P, Dusitanond P, Harnsomburana P, Laowittawas W, Chairangsaris P, Suwantamee J, Wongmek W, Ratanarat R, Poompichate A, Panyadilok H, Sutcharitchan N, Chuesuwan A, Oranrigsupau P, Sutthapas C, Tanprawate S, Lorsuwansiri J, Phattana N; Thai Botulism Study Group. An outbreak of botulism in Thailand: clinical manifestations and management of severe respiratory failure. Clin Infect Dis. 2006 Nov 15;43(10):1247-56. doi: 10.1086/508176. Epub 2006 Oct 16. PMID 17051488
- See also: Pubmed — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=17051488&query_hl=1&itool=pubmed_docsum